CLINICAL TRIAL: NCT04005287
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel, 24-Week, Phase 2a Study of Topical Pirenzepine (WST-057) or Placebo in Type 2 Diabetic Patients With Peripheral Neuropathy
Brief Title: A 24-Week Study of Topical Pirenzepine or Placebo in Type 2 Diabetic Patients (T2DM) With Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: WinSanTor, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WST-PZP-002
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Neuropathy; Painful Diabetic Neuropathy; Diabetic Neuropathies, Painful
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetic Neuropathies; Diabetes Mellitus | interventions — Pirenzepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- WST-057 Matching placebo 2 mL volume (Placebo Comparator)
  Interventions: Drug: Placebo Low Dose
- WST-057 Matching placebo 4mL volume (Placebo Comparator)
  Interventions: Drug: Placebo High Dose
- WST-057 (4% pirenzepine) 2mL volume (Active Comparator)
  Interventions: Drug: WST-057 (4% pirenzepine) Lose Dose 2mL
- WST-057 (4% pirenzepine) 4mL volume (Active Comparator)
  Interventions: Drug: WST-057 (4% pirenzepine) High Dose 4mL

INTERVENTIONS:
Drug: WST-057 (4% pirenzepine) Lose Dose 2mL — Topical Solution
  Arms: WST-057 (4% pirenzepine) 2mL volume
Drug: WST-057 (4% pirenzepine) High Dose 4mL — Topical Solution
  Arms: WST-057 (4% pirenzepine) 4mL volume
Drug: Placebo Low Dose — Topical Solution
  Arms: WST-057 Matching placebo 2 mL volume
Drug: Placebo High Dose — Topical Solution
  Arms: WST-057 Matching placebo 4mL volume

SUMMARY:
This is a randomized outpatient, double-blind, placebo-controlled, multiple-site study of the safety, tolerability, and exploratory efficacy of topically administered WST-057 (4% pirenzepine free base monohydrate) for 24 weeks in subjects with T2DM with peripheral neuropathy.

DETAILED DESCRIPTION:
This is a randomized outpatient, double-blind, placebo-controlled, multiple-site study of the safety, tolerability, and exploratory efficacy of topically administered WST-057 (4% pirenzepine free base monohydrate) for 24 weeks in subjects with T2DM with peripheral neuropathy. Subjects will attend visits at screening (day -45 to -28); day 1 (baseline); weeks 2, 4, 8, 12, 16, 20, 24; and follow-up (week 26). Approximately 60 subjects with T2DM with peripheral neuropathy will be randomized to 1 of 4 treatment groups in a 1:1:4:4 ratio: placebo control 2 mL (n = 6 subjects), placebo control 4 mL (n = 6 subjects); low dose (2 mL) WST-057 (73 mg pirenzepine free base monohydrate) (n = 24 subjects); and high dose (4 mL) WST-057 (146 mg pirenzepine free base monohydrate) (n = 24 subjects), with the assumption that a total of 50 subjects will complete the study.

This study is designed with 4 periods: screening, baseline/day 1, outpatient treatment, and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T2DM (as defined by the 2013 Diabetes Canada guidelines).
2. Male and female patients in the age range of 18 to 75 years (inclusive).
3. Presence of definite diabetic neuropathy (as defined by the Toronto Consensus Guidelines) of at least 12 months duration in the lower extremities.
4. Provide written informed consent prior to entering the study or undergoing any study procedures.
5. Females should be either not of childbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and must be practicing a highly effective medically acceptable method of contraception (e.g. abstinence, or hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); or vasectomy (partner)) for at least 1 month before the screening visit and for 1 month after the last dose of study drug. If access or use of a highly effective medically acceptable method of contraception is not achievable, then a combination of barrier methods (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) is acceptable (e.g. male condom with diaphragm, male condom with cervical cap). Eligible female subjects must also have a negative serum beta-human chorionic gonadotropin (ß-hCG) at the screening visit.
6. Males must use an acceptable form of contraception (e.g., male condom with diaphragm, male condom with cervical cap, or male condom in association with spermicide)
7. Glycemic control has been optimized and has been stable for at least three months prior to randomization. Optimal glycemic control refers to the best possible diabetic control that an individual patient can attain with usual standards of care, which usually takes more than two months to establish.
8. Patients must have a screening IENF density range of no less than 1 IENF/mm and no more than 10 IENF/mm.
9. Participating subjects must be reliable, willing, and able to cooperate with all study procedures, including the following:

   * Return for study visits on the required dates
   * Be physically able to inspect calves, tops of ankles, and soles of feet for wounds, infections, or other anomalies, and be able to self-administer the investigational drug to calves and feet.
   * Be able to accurately and reliably report symptoms (including treatment-emergent signs and symptoms).
   * Take study drug as required by protocol.
10. Be on stable antidiabetic treatment (insulin, oral agents, or lifestyle) that is not anticipated to change during the course of the study, except if medically required.
11. Be on stable analgesic treatment (same medication and dose) or stable nonpharmacological pain treatment for at least 4 weeks prior to screening and remain on this stable treatment throughout the study (unless otherwise directed by a physician). Nonpharmacologic pain treatment includes the following: relaxation/hypnosis, physical or occupational therapy, counseling, etc. Episodic or periodic treatments, such as monthly injections for treatment of pain (eg, local anesthetics), will not be permitted. Topical anesthetics/analgesics such as capsaicin, topical cannabinoid (CBD) oil or extracts, lidocaine patches and compounded topical applications are also not allowed.
12. General health status must be acceptable for participation in this 24-week clinical study, with no hospitalizations for medical conditions within 12 weeks before and during screening per judgment of the Investigator. Any question regarding eligibility will be addressed with the medical monitor.
13. Fluency (oral and written) in the language in which the standardized tests will be administered.

Exclusion Criteria:

1. Lower leg IENFD at screening of <1 or >10 IENF/mm.
2. Uncontrolled glycemia
3. Proliferative retinopathy or maculopathy requiring acute treatment.
4. Requiring dialysis.
5. Impaired liver function, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal.
6. Presence of clinically significant peripheral or autonomic neuropathy that is clearly of nondiabetic origin.
7. Uncontrolled treated/untreated hypertension (systolic blood pressure [BP] ≥ 180 or diastolic BP ≥ 100 at screening).
8. Amputations of lower extremities or presence of foot ulcers.
9. Clinically significant active macrovascular disease, including myocardial infarction or cerebrovascular event within the past 12 months.
10. Uncontrolled or untreated hypothyroidism.
11. Active infection (eg, HIV, hepatitis), or a history of severe infection during the 30 days prior to screening.
12. Evidence of severely immunocompromised status.
13. Major surgical procedure during the 90 days prior to screening.
14. Diagnosis and/or treatment of malignancy (except for basal cell or squamous cell skin cancer, in-situ carcinoma of the cervix, or in-situ prostate cancer) within the past 5 years.
15. Clinically significant gastric emptying abnormality (eg, severe gastroparesis).
16. Urinary retention or an enlarged prostate.
17. Uncontrolled glaucoma.
18. Other clinically significant, active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary, endocrine, rheumatologic or hematological system that, in the opinion of the Investigator, would compromise the subject's participation in the study, might confound the results of the study, or pose additional risk in administering the study drug.
19. New treatment with (< 3 months) antioxidant supplements, vitamins, or drugs known to affect oxidative stress and peripheral diabetic neuropathy such as Superoxide Dismutase, Alpha Lipoic Acid, Acetyl L-Carnitine and Vitamin B12.
20. Known or suspected history of alcohol or substance abuse. Moderate and stable consumption of alcohol, cannabis and nicotine are not exclusionary
21. Mental incapacity, unwillingness, or language barrier precluding adequate understanding of or cooperation with the study.
22. Women of childbearing potential who are pregnant, breast-feeding, or intend to become pregnant. Women of childbearing potential must have a negative pregnancy test at Screening and must agree to use adequate contraceptive methods during the study and for 1 month after the last dose of study drug (see inclusion criterion 5).
23. History of allergy or sensitivity to M1 antagonists or anticholinergics in general or any of the components of the investigational product formulations.
24. Known allergy or hypersensitivity to pirenzepine or another component of the investigational product.
25. History of sensitive skin, as defined by a requirement to use soap and skin products formulated for "sensitive skin".
26. Currently taking any medicines to treat overactive bladder (anticholinergic agents, such as Gelnique).
27. Failure or inability to perform screening or baseline assessments.
28. Patients with any condition that could potentially interfere with the conduct of the study or confound efficacy evaluations, including the following as specified in numbers 29 through 35 below:
29. Pain or neuropathy from another cause (as determined by the investigator) (including central pain, radiculopathy, painful arthritis, autoimmune and inflammatory diseases including rheumatoid arthritis, lupus, Sjogren's syndrome, vasculitic disorders such as periarteritis nodosa, Churg-Strauss, etc., celiac disease, Crohn's disease, ulcerative colitis, spondyloarthropathies, sarcoidosis, etc.).
30. Skin or soft-tissue lesions in the area affected by neuropathy that are painful or could alter sensation.
31. Systemic infections (eg, HIV, hepatitis, tuberculosis, syphilis).
32. Exposure to an experimental drug, experimental biologic, or experimental medical device within 3 months before screening.
33. Any open wound(s) and/or sunburn(s) in the dosing area. Subjects who have a wound and/or sunburn at screening that is anticipated to resolve before day -1 can be enrolled.
34. History of a serious skin disease (as determined by the Investigator), such as skin cancer, psoriasis, eczema or stasis dermatitis.
35. Receipt of a tattoo in the dosing area within 12 months of dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by hematology and clinical pathology blood tests. | 24 weeks
  Safety will be assessed by observing changes in patient's blood tests when compared to normal lab values/ranges after once daily dosing of 2 dose levels of WST-057 solution or placebo. The Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by vital signs (blood pressure (diastolic and systolic mmHg), heart rate (beats per minute), respiratory rate (breaths per minute). | 24 weeks
  Safety will be assessed by observing changes in vitals signs (from baseline) in patients after daily topical doses of either 2 dose levels of WST-057 solution or placebo. The Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by ECG ( measuring P Wave, QRS complex, QT Interval) | 24 weeks
  Safety will be assessed by observing changes in ECG parameters (from baseline) in patients after daily dosing of either 2 dose levels of WST-057 solution or placebo. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 will be reported.
Incidence and Treatment-Emergent Adverse Events as assessed by a dermal assessment (Draize score (scale 0.0 - 4.0) score of skin erythema, edema, pruritus and dryness score) of the dosing area | 24 weeks
  Dermal safety will be assessed by observing changes in dermal scores (from baseline) in patients after daily dosing of either 2 dose levels of WST-057 solution or placebo. The Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 will be reported.

SECONDARY OUTCOMES:
Intraepidermal Nerve Fiber Density (IENFD) | 24 weeks
  Evaluate the efficacy of WST-057 to increase IENFD present in punch biopsies collected in the calf. The nerves will be counted in these punch biopsies and the change in the density will be measured between screening and the week 24 visit. The more nerves or a higher nerve density correlates with better sensation.
Norfolk Quality of Life Measure (QOL) Patient Questionnaire | 24 Weeks
  Determine the impact of once-daily topical dosing of WST-057 on a QOL measurement. The score from the QOL questionnaire will be tabulated from each visit to determine if an improvement in the quality of life could be measured using this scale between screening and the week 24 visit.All symptoms (1-7) are scored as either a 1 or a 0, indicating a presence or absence of the symptom. With the exception of Questions 31, and 32, the other items are scored according to the 5-point Likert Scale (0-4, "No Problem" to "Severe Problem"). In Question 31, "Good", the middle item, is scored as O. "Very Good" is scored as -1, Excellent" is scored as -2. "Fair is scored as 1, and "Poor" is scored as 2. In Question 32, "About the Same", the middle item, is scored as 0. "Somewhat better" is scored as -1, "Much better" is scored as -2. "Somewhat worse" is scored as 1, and "Much worse" is scored as 2. A higher score indicates worse neuropathy-related quality of life score than a lower number.

OTHER OUTCOMES:
Quantitative Thermal Threshold (QST) Quantitative Vibration Threshold (QVT) | 24 weeks
  Determine the impact of once daily dosing of WST-057 on QST and QVT. Sensory and vibration probes attached to an instrument that measures response will be applied to the feet of patients to determine if there is an improvement from the screening visit until 24 weeks post dosing. The lower the threshold for thermal and vibration sensation indicates better feeling or less neuropathy.
Pain Assessment Scale: Visual Analogue Score | 24 weeks
  Determine the impact of once-daily topical dosing of WST-057 on the level of pain. Scores are based on self-reported measures of symptoms that are recorded with a single mark placed at one point along the length of a line that represents a continuum between the two ends of the scale-"no pain" on the left end of the scale and the "worst pain" on the right end of the scale.
Patients' Global Impression of Change | 24 weeks
  Determine the impact of once-daily topical dosing of WST-057 on the patients' perception of changes (i.e., "feeling better" or "feeling worse"). The PGIC is a 7-point verbal scale.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hansen, Study Director — WinSanTor, Inc
Locations (5):
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
  - Ottawa Hospital Research Institute Civic Campus, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CRCHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sivadasan A, Fernyhough P, Calcutt NA, Frizzi KE, Gardner K, Hansen A, Breiner A, Zochodne DW, McInnes N, Punthakee Z, Gosselin S, Perkins BA, Bril V. Topical application of the antimuscarinic pirenzepine increased lower limb nerve fibre density in a phase 2a study in type 2 patients with diabetes with peripheral neuropathy. EBioMedicine. 2026 Jan;123:106055. doi: 10.1016/j.ebiom.2025.106055. Epub 2025 Dec 5. PMID 41352124